CLINICAL TRIAL: NCT02511418
Title: Renal Hemodynamic Effects of the HMG-CoA Reductase Inhibitors in Normal Volunteers and in Patients With Chronic Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fernando Fervenza, M.D., Ph.D, Mayo Clinic
Purpose: Treatment
Other Study IDs: 475-01
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hyperlipidemia; Hypertension; Chronic Renal Failure
MeSH Terms: conditions — Hyperlipidemias; Hypertension; Kidney Failure, Chronic | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatin

SUMMARY:
This study was done to determine whether Simvastatin (a medication commonly used to treat patients with high cholesterol levels in the blood increases blood flow to the kidneys and improves renal function in normal volunteers and patients with impaired renal function secondary to polycystic kidney diseases.

ELIGIBILITY:
Patients with chronic renal failure:

1. Age 18 or older
2. Chronic renal failure secondary to Autosomal Dominant Polycystic Kidney Disease
3. Serum creatinine ≥ 1.4 but ≤ 2.0 mg/dl
4. Creatinine or iothalamate clearance between 35-70 ml/min per 1.73m2
5. Stable renal function for the three preceding months
6. Blood pressure needs to be adequately controlled (< 140/90 mm Hg), with or without the use of antihypertensive agents. However, ACE inhibitors or AT1 receptor blockers must not be initiated, or have their dose increased during the study period.

Patients with normal renal function:

1. Age 18 or older
2. Normal renal function and diagnosed with Autosomal Dominant Polycystic Kidney Disease
3. Serum creatinine ≤ 1.4
4. Creatinine or iothalamate clearance ≥70 ml/min per 1.73m2
5. Renal function has to be stable for the three preceding months
6. Blood pressure needs to be adequately controlled (< 140/90 mm Hg), with or without the use of antihypertensive agents. However, ACE inhibitors or AT1 receptor blockers must not be initiated, or have their dose increased during the study period.

Exclusion criteria include:

1. Patients using corticosteroids, cytotoxic drugs (alkylating agents, chlorambucil, cyclophosphamide), CellCept, or cyclosporin A therapy
2. Positive hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab)
3. Serum transaminase levels (AST, ALT) 2 times the upper limit of normal
4. Clinically significant medical conditions
5. Pregnant patients, patients who are breast-feeding, or women intending to conceive during the course of the study
6. Presence or suspicion of active infection, recent serious infection or chronic/recurrent viral or bacterial infection
7. Presence of concomitant renal artery stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Effect of short term HMG-CoA reductase treatment | 4 weeks
  Differences between mean values for RPF, GFR and FF at baseline versus mean values obtained for these same parameters after 4 weeks of treatment will be analyzed using two-tailed Student's paired t-test. A similar analysis will be performed regarding patient's profiles for creatinine clearance, serum creatinine, urinary protein excretion and serum lipids. All results will be expressed as mean ± standard deviations. Differences will be considered significant at P <0.05.

REFERENCES:
- [Derived] Zand L, Torres VE, Larson TS, King BF, Sethi S, Bergstralh EJ, Angioi A, Fervenza FC. Renal hemodynamic effects of the HMG-CoA reductase inhibitors in autosomal dominant polycystic kidney disease. Nephrol Dial Transplant. 2016 Aug;31(8):1290-5. doi: 10.1093/ndt/gfv394. Epub 2015 Nov 27. PMID 26614268